CLINICAL TRIAL: NCT00414284
Title: Evaluation of the Pharmacokinetics and Tolerability of Increased Dosage of Lopinavir/Ritonavir(LPV/r) in Individuals Experiencing Viremia on Standard Dose LPV/r Using LPV/r Tablet Formulation
Brief Title: BOOST: Study of Increased Dosage of Lopinavir/Ritonavir (LPV/r)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: One subject's HIV RNA rebounded at week 12. A repeat PhenoSense GT combination resistance assay at week 12 revealed evolution in protease inhibitor resistance.
Sponsor: Community Research Initiative of New England (Other)
Collaborators: Abbott (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-124; IND #71128
Record Dates: First submitted 2006-12-20; First posted 2006-12-21 (Estimated); Last update posted 2010-12-08 (Estimated); Status verified 2010-12

CONDITIONS: HIV Infections
Keywords: HIV/AIDS; viremia; Kaletra; pharmacokinetics; viral load; LPV/r; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Viremia

INTERVENTIONS:
Drug: Increased dose of Kaletra

SUMMARY:
This study will look to see if increasing the standard dose of Kaletra is tolerated and if it will lower viral loads to undetectable levels. This study will also look at the pharmacokinetic data (amount of Kaletra in blood at different times).

DETAILED DESCRIPTION:
There are several reasons for low level viremia in patients on Kaletra (LPV/r), including poor adherence, incomplete absorption, cellular drug pumps or resistance mutations. Increasing exposure to protease inhibitors via boosting with ritonavir increases minimum blood concentrations, and is a strategy which has been shown to improve suppression of virologic replication. Little is known about the pharmacokinetics (PK), tolerability and safety of increased doses of LPV/r. The objectives of this 24-week single arm pilot study are to assess the PK parameters, safety, tolerability, change in viral load and CD4 counts on increased dose (600/150 and 800/200 mg) LPV/r in participants with low level viremia on standard dose LPV/r-based ART. Participants will undergo six PK samplings over 12 hours on standard dose LPV/r. The dose will be increased to 3 tabs (600/150) BID and blood will be sampled for PK after two weeks. If tolerated at 8 weeks, the dose will be increased to 4 tabs (800/200 mg) BID and final PK sampling will be performed after two weeks. There will be a one time, optional, optimization of background regimen of NRTIs two weeks after the first dose escalation.

Major Eligibility Criteria:

* CD4 count: > 50
* Viral load: 200-75,000 on two most recent measures
* Current treatment: > 16 weeks standard dose (400/100mg BID) LPV/r-based ART (no other PI or NNRTI allowed
* Prior treatment experience and resistance profile: Up to 20-fold resistance to LPV/r

ELIGIBILITY:
Inclusion Criteria:

* CD4 Count >50
* Viral load 200-75,000 on two most recent measures
* More than 16 weeks on standard dose Kaletra (LPV/r)
* May be initial PI regimen or prior PI usage
* Up to 50-fold resistance to LPV/r

Exclusion Criteria:

* Age < 18 years old

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2006-06; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetic parameters of higher doses of LPV/r

SECONDARY OUTCOMES:
To evaluate plasma HIV-1 RNA change after increasing the dose of LPV/r
To evaluate change in CD4 count after increased dose LPV/r
To compare the tolerability and laboratory safety profile of LPV/r 3 and 4 tablets BID

CONTACTS AND LOCATIONS:
Overall Officials: Calvin J Cohen, MD, MSc, Principal Investigator — CRI
Locations (1):
- Community Research Initiative of New England - Boston, Boston, Massachusetts, United States

REFERENCES:
- See also: Web page of CRI, the nonprofit research group sponsoring the study — http://www.crine.org/